CLINICAL TRIAL: NCT06277557
Title: Evaluation of the Effects of Virtual Reality Learning Environment on Nursing Student Non-technical Skills Development: A Quasi-Experimental Study
Brief Title: Evaluation of the Effects of Virtual Reality Learning Environment on Nursing Student Non-technical Skills Development
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: HSEARS20211229002
Record Dates: First submitted 2024-01-14; First posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2022-01

CONDITIONS: Educational Problems
Keywords: Virtual Reality; Simulation

STUDY DESIGN:
Intervention Model Description: Waitlist-control study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High fidelity Simulation (Other): conventional teaching method
  Interventions: Other: Virtual Reality

INTERVENTIONS:
Other: Virtual Reality — Virtual reality learning platform as intervention in this study

SUMMARY:
The goal of this waitlist control study is to evaluate the benefits of virtual reality teaching pedagogy to developing non-technical skills in nursing students.

The main question[s] it aims to answer are:

1. What is the relationship between VR training programs and students' situation awareness skills development?
2. What is the relationship between VR training programs and students' communication skills development?
3. What is the relationship between VR training programs and students' satisfaction/self-confidence in learning?
4. What is the relationship between the sense of presence and satisfaction/ self-confidence in learning?
5. How does the student's learning experience after VR training programs?

Participants will attend the Virtual Reality training program. Researchers will compare the use of high-fidelity simulation to see if the non-technical skills were developed.

DETAILED DESCRIPTION:
The study employed a quasi-experimental, pretest-posttest, non-equivalent waitlist control group design. First, the quantitative methods were applied to obtain numerical evidence regarding statistical trends across the experimental and waitlisted control groups.

A pretest-posttest non-equivalent waitlist control group design was employed.

Convenience sampling was adopted to recruit subjects. Participants were recruited from the students who had enrolled in the subject "Clinical Reasoning and Decision Making." They were assigned into two study groups according to the tutorial teaching schedule: the control and the experimental groups. The Control group attended the usual teaching activities: simulation followed by the intervention (VR), whereas the intervention group participated in the VR (intervention) session followed by the simulation session (control).

ELIGIBILITY:
Inclusion Criteria:

* Students studying Year 3 of the Bachelor of Science in Nursing program and enrolled in the subject "Clinical Reasoning and Decision Making"

Exclusion Criteria:

* Students diagnosed with diminished visual acuity were excluded from the study to prevent the diminished visual function from affecting the VR experience.

Ages: 18 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Situation awareness and communication skills | 1) Before the intervention and waitlist control as baseline assessment; 2) immediately after the intervention or control measures as follow up assessment
  Use the "Virtual non-technical skills (v-NOTECHS)" scale (Sevidalis et al., 2008) to measure the situation awareness
Student's self-confidence in learning | 1) Before the intervention and waitlist control as baseline assessment; 2)immediately after the intervention or control measures as follow up assessment
  Use the "Student satisfaction and self-confidence in Learning" inventory (National League for Nursing, 2005) to mesure the self-confidence in learning
Participants' sense of presence in this virtual clinical environment | Immediately after the intervention or control measures
  Use the Presence Questionnaire to measure the sense of presence

CONTACTS AND LOCATIONS:
Overall Officials: Kam Hung LAI, Principal Investigator — School of Nursing, The Hong Kong Polytechnic University
Locations (1):
- Timothy LAI, Kowloon, Hong Kong

IPD SHARING:
Plan to Share IPD: No
The study result as part of the doctoral study, and the details of the IPD will not shared.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-01): https://cdn.clinicaltrials.gov/large-docs/57/NCT06277557/Prot_SAP_000.pdf
  • Informed Consent Form (2022-01-01): https://cdn.clinicaltrials.gov/large-docs/57/NCT06277557/ICF_001.pdf